CLINICAL TRIAL: NCT05645185
Title: Characterisation of Clinical Phenotypes and Outcomes of Ma2 Patient
Acronym: CarMa2
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 820
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Autoimmune Encephalitis; Paraneoplastic Syndromes
Keywords: Neurological paraneoplastic syndrome; auto immune encephalitis; Ma2 antibody
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Paraneoplastic Syndromes | interventions — Immunologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Sera, blood, DNA, CSF collected at diagnosis time
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with Ma2 antibody: This is a non-interventional study involving biological samples. Samples are already stored in biobank repositories and collected as part of "good clinical practice" in the diagnostic process of patients with suspected autoimmune encephalitis, meaning that the standard diagnostic and therapeutic approaches will not be altered in the selected study population. Patients have already gave explicit written consent for biological specimens sampling and storage at the "Centre de Ressources Biologiques des Hospices Civils de Lyon" (CRB-HCL) (including tissue, cells or biological fluids).
  Interventions: Diagnostic Test: Diagnosis test

INTERVENTIONS:
Diagnostic Test: Diagnosis test — Tests can be used: immunofluorescence, immunodot, western blot, tests CBA on sera or CSF.

SUMMARY:
Paraneoplastic neurological syndromes (PNS) are rare complications of cancer occurring in 0.01% of cases. Their clinical, biological and radiological presentation is heterogeneous and may constitute a diagnostic challenge. Anti-Ma2 PNS are rare diseases with a guarded prognosis. They are most often associated with a seminoma-like testicular tumor but can also be associated with lung cancer. Classically, they present as limbic, diencephalic and/or brainstem encephalitis. Anti-Ma2 antibodies target intracellular receptors and are characteristic of a particular form of encephalitis. Atypical manifestations including narcolepsy-cataplexy, weight gain, sexual dysfunction and motor neuron syndrome have been described and explain the difficulty in diagnosing anti-Ma2 associated PNS. It seems interesting to better characterize the phenotypes of Ma2 patients in order to optimize the diagnosis and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Neurological disorder
* Anti-Ma2 positivity in sera or CSF
* Patient > 18 years old

Exclusion Criteria:

* Patient without clinical data
* Patient without Ma2 antibody in sera or CSF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anti-Ma2 paraneoplastic neurological syndromes with or without cancer
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Rankin score | 12 month after diagnosis
  Follow up and survival (rankin score)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites autoimmunes, Lyon, France